CLINICAL TRIAL: NCT04263545
Title: A Randomised Feasibility Study Comparing a Novel Intervention for Smoking Cessation in NHS Staff to Standard Care
Brief Title: The Staff Stop Smoking Project
Acronym: STOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PHT/2019/17
Record Dates: First submitted 2020-01-29; First posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-01

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: meeting with a smoking cessation counsellor to discuss their individual requirements for smoking cessation and be offered their choice of pharmacological intervention. They will be provided with their choice of pharmacotherapy on site.They will then be invited to attend a group session, where they will have some brief lung function tests and check carbon monoxide levels. Participants will be offered refreshments and receive a bespoke group session to address various aspects of smoking cessation.
Masking Description: Participants who are randomised to the standard care arm will receive very brief advice (VBA) and signposting to local organisations to support a quit smoking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator)
  Interventions: Behavioral: Group session with smoking cessation counsellor
- Standard Care (Placebo Comparator)
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Group session with smoking cessation counsellor — Group session with smoking cessation counsellor
  Arms: Intervention
Behavioral: Standard Care — standard care arm will receive very brief advice (VBA) and signposting to local organisations to support a quit.
  Arms: Standard Care

SUMMARY:
Participants will be randomised to either standard care or to receive our help to quit programme. The study will only be available to Portsmouth Hospital Trust staff member.

DETAILED DESCRIPTION:
A randomised controlled feasibility study to trial a novel intervention to help NHS staff stop smoking compared to standard care. Participants will attend one-on-one interviews and a support group where they will undertake CO monitoring and mini-spirometry. They will complete questionnaires about their quality of life, other health problems and their general state of health. They will attend the support groups on a weekly basis and have access to support outside of these times.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, aged 18 years or over
* Willing and able to give informed consent for participation in the study.
* Must work for PHT at QAH and be able to attend weekly meetings for the duration of the study period
* Must be a current smoker

Exclusion Criteria:

-Unable to comprehend the study and provide informed consent e.g. insufficient command of English in the absence of someone to adequately interpret.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-06-21 (Actual)

PRIMARY OUTCOMES:
Behavioural outcomes | 4 weeks
  Number of smokers who achieve a successful quit
Behavioural outcomes | 12 weeks
  Number of smokers who achieve a successful quit
Behavioural outcomes | 6 months
  Number of smokers who achieve a successful quit

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Portsmouth Hospitals NHS Trust, Queen Alexandra Hospital, Portsmouth, Hampshire
  - Portsmouth Hospitals NHS Trust, Portsmouth

IPD SHARING:
Plan to Share IPD: No